CLINICAL TRIAL: NCT01204411
Title: Efficacy of the Artesunate-amodiaquine Combination for Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Between 6 and 59 Months of Age With Severe Acute Malnutrition in Madaoua, Tahoua Region, Niger
Brief Title: Efficacy of Artesunate-amodiaquine (AS-AQ) in Children With Malaria and Severe Acute Malnutrition, Madaoua, Niger 2010
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The ethics committee did not approve the pharmacokinetic part of the study.
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Spain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epicentre/Nig/2010/PaluMadaua
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Malaria, Falciparum; Malnutrition; Child
Keywords: Efficacy; Safety; Artesunate-amodiaquine; Malaria; Plasmodium falciparum; Malnutrition
MeSH Terms: conditions — Malaria, Falciparum; Malnutrition; Malaria | interventions — amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Artesunate-amodiaquine fixed-dose combination — * artesunate 25 mg / amodiaquine 67.5 mg: 1 tablet / day for 3 days for children with a weight of 5 kg to less than 9 kg;
  * artesunate 50 mg / amodiaquine 135 mg: 1 tablet / day for 3 days for children with a weight of 9 kg to less than 18 kg;
  * artesunate 100 mg / amodiaquine 270 mg: 1 tablet / day for 3 days for children with a weight of 18 kg to less than 36 kg;
  Other Names: AS-AQ Winthrop® Sanofi Aventis

SUMMARY:
The purpose of the study is to determine whether the artesunate-amodiaquine combination is effective in treating uncomplicated Plasmodium falciparum malaria in children with severe acute malnutrition.

Infection with Plasmodium falciparum malaria remains a significant cause of morbidity and mortality in malnourished children. Malnutrition is known to have a modulating effect on the incidence of malaria infections, its severity and effectiveness of treatments. However, little data exists on antimalarial drug efficacy in malnourished children. Artesunate-amodiaquine combination is the first line treatment used in Médecins Sans Frontières programmes in Niger. The assumption of current efficacy of artesunate-amodiaquine is based on non malnourished children. The aim of this study is to measure the clinical and parasitological efficacy in severely malnourished children.

The study is consistent with the standard WHO protocol for monitoring antimalarial drug efficacy (WHO: Methods for surveillance of antimalarial drug efficacy. Geneva; 2009), except for one inclusion criterion. Severe acute malnutrition is an inclusion criteria, instead of being an exclusion criteria. The study will encompass a pharmacokinetic part that will provide important information on the absorption of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 59 months
* Weight ≥5kg
* P. falciparum monoinfection confirmed on a thick blood film
* Parasitic density between 1,000 and 200,000 asexual forms/uL of blood
* Measured axillary temperature ≥37.5°C or history of fever during the previous 24 hours
* Severe malnutrition (defined as a weight/height ratio less than -3 z-scores)
* High probability of compliance with follow-up visits (home is within two hours of walk from the outpatient department, no near-term travel plans, etc..)
* Consent of a parent or guardian who is at least 18 years of age.

Exclusion Criteria:

* Signs of a critical illness as defined by the WHO (WHO (2000) Severe falciparum malaria; Clinical features of severe falciparum malaria in children. Royal Society of Tropical Medicine and Hygiene, 94 (supplement 1), 5-11).
* Signs of severe or complicated malaria as defined by the WHO (WHO (2000) Severe falciparum malaria; Clinical features of severe falciparum malaria in children. Royal Society of Tropical Medicine and Hygiene, 94 (supplement 1), 5-11).
* Severe anaemia (haemoglobin <5 g/dL)
* Known history of hypersensitivity to any of the study medications,
* Symmetric oedema in the feet,
* Concomitant febrile illness not originating from malaria, which could alter the outcome of the study (measles, acute lower respiratory tract infection, otitis media, tonsillitis, abscesses, severe diarrhea with dehydration, etc.),
* History of a full treatment course with the study drug in the past 28 days.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To measure the PCR adjusted clinical and parasitological efficacy of the artesunate-amodiaquine combination in children 6-59 months of age with severe malnutrition and uncomplicated P. falciparum malaria over a period of 42 days. | 42 day follow-up

SECONDARY OUTCOMES:
To assess the incidence of adverse events during the follow-up period | 42 day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Grandesso, MSc, Principal Investigator — Epicentre
Locations (1):
- Integrated health centre (CSI), Madaoua, Tahoua Region, Niger